CLINICAL TRIAL: NCT05340816
Title: The Effect of Manual Lymphatic Drainage and Transcutaneous Electrical Nerve Stimulation Methods in Women with Premenstrual Syndrome
Brief Title: The Effects of Manual Lymphatic Drainage and Transcutaneous Electrical Nerve Stimulation in Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Gamze Kurt, associate professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMS-1
Record Dates: First submitted 2022-04-06; First posted 2022-04-22 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Premenstrual Syndrome
Keywords: Manual Lymphatic Drainage; Transcutaneous Electrical Nerve Stimulation; Premenstrual Syndrome; Quality of Life; Autonomic Functions
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Manual Lymphatic Drainage; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to manual lymph drainage, transcutaneous electrical nerve stimulation, or a control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The researcher who made the assessments and participants do not know which group participants belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Manual Lymphatic Drainage (Experimental): 5 days, 30 minutes, Manual Lymphatic Drainage
  Interventions: Other: Manual Lymphatic Drainage
- Transcutaneous Electrical Nerve Stimulation (Experimental): 5 days, 20 minutes, Transcutaneous Electrical Nerve Stimulation
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- Control (No Intervention): no any intervention

INTERVENTIONS:
Other: Manual Lymphatic Drainage — Manual lymphatic drainage will apply to the neck, abdominal, bilateral inguinal lymph nodes, bilateral anterior/posterior thighs, and lumbal area. Treatment duration will be approximately 30 minutes for 5 days.
  Arms: Manual Lymphatic Drainage
Device: Transcutaneous Electrical Nerve Stimulation — Transcutaneous electrical nerve stimulation will be apply to abdominal and lumbal area as 100 Hz and 100 msn. Treatment duration will be approximately 20 minutes for 5 days.
  Arms: Transcutaneous Electrical Nerve Stimulation

SUMMARY:
The aim of this study is to (a) investigate the effects of manual lymphatic drainage and transcutaneous electrical nerve stimulation on the severity of syndrome symptoms, pain, heart rate variability, and quality of life in women with premenstrual syndrome, and (b) compare the effectiveness of these two methods. Female participants who met the inclusion criteria and volunteered to participate in the study will be called approximately one week before menstruation. After the participants are randomly divided into 3 groups, their baseline assessments will be made. Then, the participants will be treated according to the group they are assigned to. Treatments will be applied for 5 days and once a day. No treatment will be applied to the control group. The assessments will be repeated after the treatment, on 1st day of menstruation, two days before the next menstruation, and on the first day of the next menstruation. The hypothesis of this study is that manual lymphatic drainage and transcutaneous electrical nerve stimulation have positive effects on the severity of premenstrual syndrome symptoms, pain, heart rate variability, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* women aged between18-45 years-old
* regular menstrual cycles (cycles of 21-35 days with a bleeding time of 3-10 days)
* premenstrual syndrome (according to the premenstrual syndrome scale, be above 110 points)

Exclusion Criteria:

* pregnancy
* premenstrual dysphoric disorder
* menopause
* chronic disease
* continuous use of medication
* under hormonal therapy
* infection
* using any method to cope with premenstrual syndrome

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
The Premenstrual Syndrome Scale (PMSS) | 1 month
  PMSS will be used to measure the severity of premenstrual symptoms. The participant is asked to mark retrospectively, taking into account the "being within the period one week before the menstrual period". There are 44 items in the scale. The scale items have a five-point Likert type rating ranging from 1 to 5. The lowest score that can be obtained from the scale is 44, and the highest score is 220. A higher PMSS score indicates more severe premenstrual symptoms.

SECONDARY OUTCOMES:
Heart rate and Heart rate variability | 1 month
  Heart rate (HR) is the speed of the heartbeat measured by the number of contractions (beats) of the heart per minute. Heart rate variability (HRV) is the physiological phenomenon of variation in the time interval between heartbeats. It is measured by the variation in the beat-to-beat interval. A heart rate sensor will be used to evaluate HR and HRV.
Visual analog scale (VAS) for pain levels | 1 month
  The VAS will use to assess the participants' pain levels. In the VAS, patients are asked to mark the severity of their pain on a scale from 0 to 10. The VAS ranges from '0' representing no pain and '10' representing the worst pain.
Short form of the World Health Organization Quality of Life Questionnaire (WHOQOL) | 1 month
  WHOQOL will be used to assess quality of life.WHOQOL-BREF consists of four sub-dimensions (physical health, psychological health, social relations, and environment) and a total of 27 questions. Participants are asked to answer considering the last 15 days. Each question is scored between 1 and 5, and higher scores on the sub-dimensions indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze KURT, Ph.D., Principal Investigator — Kutahya Health Science University
Locations (1):
- Kutahya Health Sciences University- Health Sciences Faculty, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohebbi Dehnavi Z, Jafarnejad F, Sadeghi Goghary S. The effect of 8 weeks aerobic exercise on severity of physical symptoms of premenstrual syndrome: a clinical trial study. BMC Womens Health. 2018 May 31;18(1):80. doi: 10.1186/s12905-018-0565-5. PMID 29855308
- [Background] Heydari N, Abootalebi M, Jamalimoghadam N, Kasraeian M, Emamghoreishi M, Akbarzadeh M. Investigation of the effect of aromatherapy with Citrus aurantium blossom essential oil on premenstrual syndrome in university students: A clinical trial study. Complement Ther Clin Pract. 2018 Aug;32:1-5. doi: 10.1016/j.ctcp.2018.04.006. Epub 2018 Apr 14. PMID 30057033
- [Background] Ghaffarilaleh G, Ghaffarilaleh V, Sanamno Z, Kamalifard M. Yoga positively affected depression and blood pressure in women with premenstrual syndrome in a randomized controlled clinical trial. Complement Ther Clin Pract. 2019 Feb;34:87-92. doi: 10.1016/j.ctcp.2018.11.007. Epub 2018 Nov 9. PMID 30712751